CLINICAL TRIAL: NCT04096898
Title: Clinical Trial to Determine Whether Senofilcon A Lenses Provide Relief of Symptoms and Signs in Patients With Moderate to Severe Dry Eye Disease
Brief Title: Senofilcon A Lenses in Moderate to Severe Dry Eye Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Principal Investigator, Timothy T. McMahon, OD, Dr. Timothy T. McMahon, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-0941
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Moderate to Severe Dry Eye Disease
Keywords: dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Senofilcon A contact lens — Senofilcon lenses will be tested in moderate to severe dry eye patients to determine their efficacy in reducing discomfort associated with dry eye.

SUMMARY:
A clinical trial using Senofilcon A daily lenses in the treatment of moderate to severe dry eye. This a comparison between signs and symptoms prior to and during treatment.

DETAILED DESCRIPTION:
32 patients with moderate to severe dry eye will be enrolled in this short-term proof of concept study to determine the efficacy in using soft lenses made of Senofilcon A in reducing signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of moderate to severe dry eye associated with either Graft-versus-host disease (GVHD), Sjogren syndrome, idiopathic dry eyes, or minimal limbal cell deficiency
* A baseline Schirmer tear test (1) of less than 5 mm at 5 minutes without anesthesia
* Have a visual analog score for comfort of 50 or less (scale of 1-100, with 100 meaning perfect ocular comfort and 1 meaning severe ocular pain)
* Ability or the resources to insert and remove the study lenses
* An OSDI score greater than 42
* A willingness to sign an informed consent

Exclusion Criteria:

* No dry eyes or mild dry eyes
* A baseline Schirmer tear test (1) of greater than 5 mm of wetting at 5 minutes
* Dry eye comfort score of greater than 50 on a visual analog scale
* Unable to insert or remove the study lenses (or have a family member do so)
* Have an OSDI score less than 42
* Has been diagnosed with neurotrophic keratopathy in either eye
* Unwilling to enroll in the study, and unwilling to provide signed informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | 2 weeks
  Patient questionaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided